CLINICAL TRIAL: NCT03763253
Title: Local Cytoreductive Treatments for Men With Newly Diagnosed Metastatic Prostate Cancer in Addition to Standard of Care Treatment
Brief Title: Additional Treatments to the Local Tumour for Metastatic Prostate Cancer: Assessment of Novel Treatment Algorithms
Acronym: IP2-ATLANTA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 18HH4804
Record Dates: First submitted 2018-11-12; First posted 2018-12-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care; Prostatectomy; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Three-arm unblinded randomised controlled trial using a positive control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm: Standard of Care (SOC) (Active Comparator): Standard of Care (SOC) treatment as determined by treating physician (positive control) (androgen deprivation with or without docetaxel chemotherapy or other systemic standard of care treatment including but not limited to Abiraterone or Enzalutamide).
  Radiotherapy to the prostate in this arm is defined as cytoreductive (for symptom control) in high volume (>/=4) metastases or to mirror current accepted local radiotherapy dose regimens for men with low volume metastases (<4 metastases).
  Metastases directed therapy will not be permitted in the control arm. Palliative radiotherapy for symptom control or for prevention of fracture will be permitted as standard clinical practice.
  Interventions: Combination Product: Standard of Care
- Intervention Arm 1: Minimally Invasive Ablative Therapy (MIAT) (Active Comparator): MIAT to prostate in form of cryotherapy or high intensity focused ultrasound (HIFU), in addition to SOC systemic treatment. No local prostate radiotherapy will be given as part of this intervention. Radiotherapy can be given subsequently for palliative reasons.
  Metastatic directed therapy will be available for use in this arm (if declared at randomisation).
  Interventions: Combination Product: Standard of Care; Procedure: Minimally Invasive Ablative Therapy (MIAT)
- Intervention Arm 2: Radical Therapy (Active Comparator): Radical therapy in form of prostatectomy (any approach) or external beam radiotherapy (radical dose) in addition to SOC systemic treatment. Modality based on physician and patient preference and patient co-morbidities.
  For patients undergoing radical prostatectomy no local prostate radiotherapy will be given as part of the intervention. Radiotherapy can be given subsequently for palliative reasons.
  Radical radiotherapy doses in this arm will be higher than SOC.
  Metastatic directed therapy will be available for use in this arm (if declared at randomisation).
  Interventions: Combination Product: Standard of Care; Procedure: Radical Therapy (Prostatectomy or Radiotherapy)

INTERVENTIONS:
Combination Product: Standard of Care — Androgen deprivation with or without docetaxel chemotherapy, Abiraterone, Enzalutamide or any other proven agent) treatment as determined by treating physician (positive control).
Procedure: Minimally Invasive Ablative Therapy (MIAT) — MIAT includes High intensity focused ultrasound (HIFU) or Cryotherapy to the prostate.
  Metastatic Directed Therapy available for use.
  Other Names: Metastatic Directed Therapy (MDT)
  Arms: Intervention Arm 1: Minimally Invasive Ablative Therapy (MIAT)
Procedure: Radical Therapy (Prostatectomy or Radiotherapy) — Radical therapy includes: Prostatectomy (any surgical approach) or External beam radiotherapy (High dose).
  Metastatic Directed Therapy available for use.
  Other Names: Metastatic Directed Therapy (MDT)
  Arms: Intervention Arm 2: Radical Therapy

SUMMARY:
Local cytoreductive treatments for men with newly diagnosed metastatic prostate cancer in addition to standard of care treatment

DETAILED DESCRIPTION:
TITLE: Additional Treatments to the Local tumour for metastatic prostate cancer: Assessment of Novel Treatment Algorithms (ATLANTA)

OBJECTIVES: To determine whether the addition of local treatment to the prostate (minimally invasive therapy or radical therapy [prostatectomy or radiotherapy]), including selective metastases-directed therapy, improves oncological outcomes in men receiving standard of care treatment for newly diagnosed metastatic prostate cancer

PHASE: Phase II Randomised Control Trial (RCT) incorporating an internal pilot

DESIGN: Three-arm unblinded randomised controlled trial using a positive control

SAMPLE SIZE: 432

POPULATION: Men who are willing to undergo local therapy to the prostate and selective metastases-directed therapy for metastatic prostate cancer in addition to standard care systemic treatment.

STUDY HYPOTHESIS: We hypothesise that men with metastatic disease who undergo treatment of the local tumour in the form of either radical therapy (prostatectomy or radiotherapy) or minimally invasive ablative therapy (MIAT), combined with metastases directly therapy, will have improved survival compared to those who receive standard of treatment alone. We will be investigating this newly evolving treatment paradigm in a formal randomised control trial (RCT).

TREATMENT/MAIN STUDY PROCEDURES: (including treatment duration and follow-up) Our pragmatic design ensures all eligible patients can be approached and randomised as there is no requirement for fitness to undergo RP. The design also incorporates the latest approach for standard of care as well as management of lymph nodes.

Arm 1*: Standard of Care (SOC) treatment as determined by treating physician (positive control) (androgen deprivation with or without Docetaxel chemotherapy or other systemic/local directed standard of care treatment including but not limited to Abiraterone or Enzalutamide). Radiotherapy in this arm defined as palliative/cytoreductive in high volume metastases or to mirror STAMPEDE local radiotherapy arm in low volume metastases.

Arm 2**: Minimally Invasive Ablative Therapy (MIAT) to local tumour / prostate in addition to SOC systemic treatment. Predominantly cryotherapy but based on disease characteristics, HIFU also. Metastases directed therapy declared prior to randomisation.

Arm 3**: Radical therapy (Prostatectomy or External beam radiotherapy [60Gy x 20 or 74Gy + in 32-37 weeks]) in addition to SOC systemic treatment. Modality based on physician and patient preference and patient co-morbidities. Metastases directed therapy declared prior to randomisation.

FOLLOW-UP DURATION: Until progression or minimum 2-years or maximum 4 years whichever is first (or 6 months for the Pilot if the trial does not progress to Phase II).

Prior to enrolment all patients must undergo Standard of Care (SOC) staging investigations for localised and metastatic disease and will need to have histologically proven local disease within the prostate. There will be no restriction on the type of biopsy used for diagnosis.

*ADT but not chemotherapy may be initiated prior to recruitment.The decision as to which SOC systemic therapy regimen will be used is by the treating clinician and/or clinical team (to be declared upfront prior to randomisation). If radiotherapy is planned for local disease in some cases in the SOC arm then this will be declared upfront prior to randomisation by the treating physician. Similarly, if lymph node radiotherapy is to be advocated then this is to be declared upfront prior to randomisation by the treating physician and can be applied to any one of the three arms. Randomisation into a treatment arm would occur at the time of recruitment which would be within 3 months of starting SOC systemic therapy.

Extra blood and urine samples will be identified using a special study number assigned to each patient, in such a way that the scientists analysing them will not be able to find out patients identity.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with prostate cancer within 6 months of screening visit
2. Metastatic disease (Any T, Any N, M1+) of any grade, stage or Prostate Specific Antigen (PSA) level.
3. Fit to undergo standard of care treatment for metastatic disease and both minimally invasive therapy and prostate radiotherapy/prostatectomy.
4. Performance status 0-2
5. Histologically proven local tumour

Exclusion Criteria:

1. Patient did not undergo and/or is unable to undergo standard of care baseline imaging tests for confirmation of metastatic status (CT abdomen/pelvis AND chest Xray (or CT chest) AND radioisotope bone scan (or whole body imaging such as MRI or PET imaging as alternative to all preceding scans mentioned here) AND prostate MRI.
2. Prior exposure to long-term androgen deprivation therapy or hormonal therapy for the treatment of prostate cancer unless started within 6 months of screening visit.
3. Prior chemotherapy or local or systemic therapy for treatment of prostate cancer (apart from ADT or hormonal therapy as outlined above)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 433 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Prostate cancer on post-standard of care prostate biopsy. | 6 months
  Proportion of patients with complete pathological response, measured on post SOC (systemic therapy) prostate biopsies (Internal Pilot).
Safety (Adverse Events) | 2-4 years (continuous)
  Safety (Adverse Events), measured using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0, Grade 1-5.
Progression-free survival (PFS) | 2-4 years
  Progression-free survival (PFS), measured as a composite outcome of Biochemical failure (PSA progression value) or Local progression or Lymph node progression or Bone metastases progression (new sites) or Progression or development of new distant metastases, defined as lymph nodes outside the pelvis, bone or organ involvement or Skeletal-related events confirmed as progression as in the Systemic Therapy in Advancing Or Metastatic Prostate Cancer: Evaluation Of Drug Efficacy (STAMPEDE) RCT).

SECONDARY OUTCOMES:
Urinary side effects | Baseline, week 26, 52, then at 24 months.
  Urinary side effects, measured using the IPSS questionnaire, Score 0-35.
Sexual side effects | Baseline, week 26, 52, then at 24 months.
  Sexual side effects, measured using the IIEF15 questionnaire, Score 0-75.
Rectal side effects | Baseline, week 26, 52, then at 24 months.
  Rectal side effects, measured using the EPIC bowel and bladder questionnaire, Score 14-113.
Progression (Biochemical / Radiological / Clinical) | Baseline, week 12, 26, 34, 52 then every every 24 weeks for remaining years 2 to 4 and Imaging tests at baseline and if progression is suspected by a clinician
  Progression on PSA and imaging and impact of clinical features on progression, measured using PSA blood tests
Health-related quality-of-life | Baseline, week 26, 52, then at 24 months.
  Health-related quality-of-life, measured using EuroQol (EQ-5D-5L) questionnaire, Score 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Hashim U Ahmed, FRCS Urol, Principal Investigator — Imperial College London
Locations (21):
- United Kingdom (21):
  - Wirral University Teaching Hospital, Wirral University Teaching Hospital NHS Foundation Trust, Birkenhead
  - Glan Clwyd Hospital, Bodelwyddan
  - Darent Valley Hospital, Dartford
  - Royal Devon and Exeter NHS Trust, Exeter
  - Buckinghamshire Healthcare NHS Trust, High Wycombe
  - West Middlesex University Hospital, Isleworth
  - Queen Elizabeth Hospital, Kings Lynn, Kings Lynn
  - Chelsea and Westminster Hospital, London
  - The Royal Marsden NHS Foundation Trust, Chelsea Research Centre, London
  - Imperial College Healthcare NHS Trust, London
  - North Middlesex University Hospital, London
  - Northwick Park, London North West Healthcare NHS Trust, London
  - St George's University Hospital, London
  - University College London Hospital, London
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Freeman Hospital, Newcastle, Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Oxford University Hospital, Oxford
  - Southampton General Hospital, University Hospital Southampton NHS Foundation Trust (UHS), Southampton
  - Sunderland Royal Hospital, City Hospitals Sunderland NHS Foundation Trust, Sunderland
  - Croydon University Hospital, Thornton Heath
  - Southend University Hospital, Westcliff-on-Sea

REFERENCES:
- [Derived] Connor MJ, Shah TT, Smigielska K, Day E, Sukumar J, Fiorentino F, Sarwar N, Gonzalez M, Falconer A, Klimowska-Nassar N, Evans M, Naismith OF, Thippu Jayaprakash K, Price D, Gayadeen S, Basak D, Horan G, McGrath J, Sheehan D, Kumar M, Ibrahim A, Brock C, Pearson RA, Anyamene N, Heath C, Shergill I, Rai B, Hellawell G, McCracken S, Khoubehi B, Mangar S, Khoo V, Dudderidge T, Staffurth JN, Winkler M, Ahmed HU. Additional Treatments to the Local tumour for metastatic prostate cancer-Assessment of Novel Treatment Algorithms (IP2-ATLANTA): protocol for a multicentre, phase II randomised controlled trial. BMJ Open. 2021 Feb 25;11(2):e042953. doi: 10.1136/bmjopen-2020-042953. PMID 33632752